CLINICAL TRIAL: NCT06493500
Title: Efficacy of Nano-hydroxyapatite Containing Tooth Paste on Dentin Hypersensitivity of Adult Patient
Brief Title: Efficacy of Formulated Eggshell Derived Nano-hydroxyapatite Containing Toothpaste With and Without Addition of Fluoride vs. Conventional Desensitizing Fluoride Containing Toothpaste in Management of Dentin Hypersensitivity
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, shahenda gamal tawfik hamdy, dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: cebc-cu-2024-06-30
Record Dates: First submitted 2024-06-30; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Dentin Hypersensitivity; Fluoride; Nano-hydroxy Apatite
MeSH Terms: conditions — Dentin Sensitivity | interventions — Toothpastes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: * This study is a double blinded study, the participants as well as the assessors will be blinded. The operator will not be blinded to apply both interventions following the manufacturer's instructions.
  * Double blinded study design is the recommended design for studies of DH. (Holland et al., 1997)
  * Outcome assessors and analyst (M.S and D.E) will be blinded to the intervention group assigned to the patients.
  * Operator (SH.G) will not be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eggshell derived Nano-hydroxyapatite (n-HAp) with Fluoride containing toothpaste (Experimental): patients would be instructed to treat their teeth for 5 min twice a day with the provided toothpaste.
  Interventions: Drug: Eggshell derived Nano-hydroxyapatite (n-HAp) with a Fluoride containing toothpaste
- Eggshell derived Nano-hydroxyapatite (n-HAp) without Fluoride containing toothpaste (Experimental): patients would be instructed totreat their teeth for 5 min twice a day with the provided toothpaste.
  Interventions: Drug: Eggshell derived Nano-hydroxyapatite (n-HAp) without a Fluoride containing toothpaste
- Commercially available Fluoride containing toothpaste (Sensodyne Rapid Relief) (Active Comparator): patients would be instructed totreat their teeth for 5 min twice a day with the provided toothpaste.
  Interventions: Drug: Eggshell derived Nano-hydroxyapatite (n-HAp) with a Fluoride containing toothpaste

INTERVENTIONS:
Drug: Eggshell derived Nano-hydroxyapatite (n-HAp) with a Fluoride containing toothpaste — patients would be instructed to treat their teeth for 5 min twice a day with the provided toothpaste.
  Other Names: (n-HAp) toothpaste
  Arms: Commercially available Fluoride containing toothpaste (Sensodyne Rapid Relief); Eggshell derived Nano-hydroxyapatite (n-HAp) with Fluoride containing toothpaste
Drug: Eggshell derived Nano-hydroxyapatite (n-HAp) without a Fluoride containing toothpaste — patients would be instructed to treat their teeth for 5 min twice a day with the provided toothpaste.
  Other Names: nano-hydroxyapatite with flouride
  Arms: Eggshell derived Nano-hydroxyapatite (n-HAp) without Fluoride containing toothpaste

SUMMARY:
compare the effectiveness of Eggshell derived nano-Hydroxyapatite with and without fluoride and conventional fluoride containing tooth paste versus conventional desensitizing fluoride containing tooth paste on dentinal tubule occlusion and dentin mineral deposition.

DETAILED DESCRIPTION:
Recently advanced nanotechnology has taken a wide leap in improving the various measures in the treatment of hypersensitivity by its nanoparticles. Nanoparticles can easily penetrate into dentin tubules, which could act as mineralizing agents that block fluid movement within the dentin tubules when combined with various agents.

Hydroxyapatite (HAp) is the major inorganic component of natural teeth and bone. Nano-sized particles of hydroxyapatite are similar to the apatite crystals of tooth enamel in morphology and crystal structure and has been studied as a biomimetic material for the reconstruction of tooth enamel suffering from mineral loss because of its unique potential for remineralization. Nano-hydroxyapatite (n-HAp) was considered a promising active ingredient used for the treatment of DH due to high biocompatibility and bioactivity. In toothpastes, HAp was included in the form of nanocrystals because they dissolve easier in this form. Crystals of n-HAp included in dental products have a dimension of 50-1000 nm, which enables them to act like fillers. These products can penetrate and block the exposed dentinal tubules which are responsible for DH

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients Aged 18-60
* Males or females.
* Good oral hygiene
* Absence of abnormal occlusion habits (e.g. bruxism, nail biting, tooth clenching and mouth breathing).
* Teeth with hypersensitivity, VAS ≥5
* Co-operative patients who show interest to participate in the study.

Exclusion Criteria:

* Patients with known allergic or adverse reaction to the tested materials.
* Systematic disease that may affect participation.
* Xerostomic patients.
* Patients with bad oral hygiene
* Patients with orthodontic appliances, or bridge work that might interfere with evaluation
* Patients who did any periodontal surgeries within the previous 6 months.
* Patients with physical disabilities

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Pain intensity due to Dentin Hypersensitivity by Visual Analogue Scale (VAS) | T (Time): T0= Baseline (before treatment). T1= 7 days. T2= 3 months. T3= 6 months
  VAS is used to "quantify" the pain severity in millimeter (mm) in response to such query as "Draw a line on the scale that shows how much pain you have at this time " with "no pain" on the far left end of scale at 0 mm and "pain as bad as it can be" on the far right at 100 mm.